CLINICAL TRIAL: NCT04330716
Title: Genetic Testing for Breast, Ovarian, Pancreatic, and Prostate Cancers - GeneBOPP
Brief Title: Genetic Testing for Breast, Ovarian, Pancreatic, and Prostate Cancers
Acronym: GeneBOPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Ambry Genetics (Industry)
Responsible Party: Principal Investigator, Huma Rana, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-652
Record Dates: First submitted 2020-03-17; First posted 2020-04-01 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Metastatic Prostate Cancer
Keywords: Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Metastatic Prostate Cancer; Genetic Counseling; Genetic Testing
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Standard genetic counseling (Active Comparator): Will receive standard genetic counseling prior to genetic testing.
  Interventions: Behavioral: Standard Genetic Counseling
- Group B: Educational video (Experimental): Will watch a brief educational video that is approximately 8 minutes in length about the genetic testing process and what to expect prior to genetic testing.
  Interventions: Behavioral: Educational Video

INTERVENTIONS:
Behavioral: Standard Genetic Counseling — Standard of care genetic counseling
  Arms: Group A: Standard genetic counseling
Behavioral: Educational Video — Video tutorial about genetic testing
  Arms: Group B: Educational video

SUMMARY:
This study is evaluating the effect of two pre-test education methods on participants interested in genetic testing for hereditary cancer risk.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial will evaluate the effect of two pre-test education methods on the level of participation in genetic testing for hereditary cancer risk. A prospective study examines outcomes before the development of a disease.

* The research study procedures include screening for eligibility, randomization and a series of questionnaires.
* Participants will be randomized, or assigned by chance, to one of two methods of pre-genetic test education and after completing either pre-test education participants will be offered the opportunity to have genetic testing performed

Two methods of pre-genetic test education:

* video education
* in-person counseling
* Genetic testing will be performed by blood draw.
* It is expected that 500 people will participate in this study
* Participants will be in the research study for up to 5 yrs after enrollment

ELIGIBILITY:
Inclusion Criteria:

* Potentially eligible participants will be identified via medical record screening and/or in accordance with their clinical visit. A HIPAA waiver of authorization will be obtained by the enrolling Institution as needed to have access to the subject's medical record information for screening of eligibility.
* A member of the study team will approach the potentially eligible participant in clinic and discuss the trial. Potentially eligible participants may choose to discuss participation further with their physician at their appointment
* Age ≥ 18 years
* Breast, ovarian, pancreatic, or metastatic prostate cancer
* No prior cancer genetic testing
* Ability to understand and the willingness to sign an informed consent document

Exclusion Criteria:

* Pregnant
* Prisoners
* Inability to understand English as a spoken language in a healthcare context
* Known hematologic malignancy (e.g. CLL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of patients who have germline genetic tests | Up to 3 years
  Measurement of genetic testing uptake in breast, ovarian, pancreatic, and prostate cancer patients randomized to pre-genetic test (pre-test) in-person counseling with a genetic counselor per standard of care or video education.This comparison will use a two-sided Fisher exact test

SECONDARY OUTCOMES:
Patient Satisfaction Survey following intervention | Immediately following intervention
  Measurement and comparison by randomized arm and communication of results of patient satisfaction using survey instruments. Administered immediately following the intervention. The survey evaluates the subject's satisfaction with the genetic testing process for both arms.
Result Disclosure Preference following intervention | Immediately following intervention
  Measurement and comparison by randomized arm and communication of results of patient disclosure preferences using survey instruments. Administered immediately following the intervention.
Patient Satisfaction 2 months following intervention | after results have been received, two months post-intervention
  Measurement and comparison by randomized arm and communication of results of patient satisfaction using survey instruments. Administered two months after the intervention. The survey evaluates the subject's satisfaction with the genetic testing process for both arms.
Psychological distress following intervention | after results have been received, two months post-intervention
  MICRA is a widely used validated 25-item measure that assesses psychosocial consequences associated with genetic testing for cancer. Section 1 contains 3 sub-scales: the Positive sub-scale (4 items), the Distress sub-scale (6 items), and the Uncertainty sub-scale (9 items) and two other items that do not fit into either sub-scale. Section 2 contains two items for participants who have children. Section 3 contains 2 items for participants who have/have had cancer. Responses are indicated on a 4 point scale for experiences in the past week. A higher score in the sub-scales or total scale indicated greater distress. The positive sub-scale is reverse scored to reflect this.
Knowledge about genetics testing | Immediately following intervention
  Measurement and comparison by randomized arm and communication of results of Patient knowledge about genetics testing using survey instruments. Knowledge about genetic testing is evaluated through a Knowledge of Multigene Panel Testing survey immediately following the intervention.
Decisional Regret | after results have been received, two months post-intervention
  Measurement and comparison by randomized arm and communication of results of Patient decisional regret to have genetic testing. Decisional regret is evaluated through a decisional regret survey that is administered two months after intervention.
Family communication of genetic test results | after results have been received, two months post-intervention
  Measurement of family communication. Family communication survey is administered two months following the intervention.
Positive Results impact | after results have been received, four months post-intervention
  Measurement of impact of positive results for patients who tested positive for a genetic mutation. This survey is administered four months post-intervention.
Cascade testing in positives | after results have been received, four months post-intervention
  Measurement of cascade testing for patients who tested positive for a genetic mutation. This survey is administered four months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Rana, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - Lifespan Cancer Institute at Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu